CLINICAL TRIAL: NCT06752005
Title: The Effects of Positioning on Comfort, Stress Levels, and Physiological Functions in Premature Infants Receiving Non-Invasive Mechanical Ventilation: A Randomized Crossover Study
Brief Title: The Effect of Positioning on Comfort, Stress Levels, and Physiological Functions in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, funda güler, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional Randomize Study
Record Dates: First submitted 2024-12-17; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Position on Premature Infants; Nursing Care
Keywords: Mechanical ventilation; Patient comfort; Nursing care; Premature infants
MeSH Terms: conditions — Premature Birth | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Following recruitment, the infants were divided into three groups, and each group was positioned in three different postures sequentially using a crossover method by randomization (1:1 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group supine, quarter prone, prone (Experimental): One of the investigators created a randomization sequence using a simple random numbers table and determined the groups. Another researcher assigned premature infants to the study groups according to the order of hospitalization in the unit, and the same researcher also applied the intervention. Thus, each infant experienced all three positions in a crossover design by the end of the study. Infants in all three groups were positioned for two hours in each posture, totaling six hours by the end of the study. Immediately after positioning in each posture, and at 1, 30, 60, 90, and 120 minutes, heart rate and oxygen saturation (SpO₂) values were recorded from bedside monitors, and respiratory rate was counted over one minute. Comfort and stress scores were assessed immediately after positioning (1 minute) and at 60 and 120 minutes. The Premature Infant Comfort Scale (PICS) was used to assess comfort, while the Neonatal Stress Scale (NSS) was used to evaluate stress.
  Interventions: Behavioral: Intervention Group
- Intervention Group quarter prone, prone, supine (Experimental): One of the investigators created a randomization sequence using a simple random numbers table and determined the groups. Another researcher assigned premature infants to the study groups according to the order of hospitalization in the unit, and the same researcher also applied the intervention. Thus, each infant experienced all three positions in a crossover design by the end of the study. Infants in all three groups were positioned for two hours in each posture, totaling six hours by the end of the study. Immediately after positioning in each posture, and at 1, 30, 60, 90, and 120 minutes, heart rate and oxygen saturation (SpO₂) values were recorded from bedside monitors, and respiratory rate was counted over one minute. Comfort and stress scores were assessed immediately after positioning (1 minute) and at 60 and 120 minutes. The Premature Infant Comfort Scale (PICS) was used to assess comfort, while the Neonatal Stress Scale (NSS) was used to evaluate stress.
  Interventions: Behavioral: Intervention Group
- Intervention Group prone, supine, quarter prone (Experimental): One of the investigators created a randomization sequence using a simple random numbers table and determined the groups. Another researcher assigned premature infants to the study groups according to the order of hospitalization in the unit, and the same researcher also applied the intervention. Thus, each infant experienced all three positions in a crossover design by the end of the study. Infants in all three groups were positioned for two hours in each posture, totaling six hours by the end of the study. Immediately after positioning in each posture, and at 1, 30, 60, 90, and 120 minutes, heart rate and oxygen saturation (SpO₂) values were recorded from bedside monitors, and respiratory rate was counted over one minute. Comfort and stress scores were assessed immediately after positioning (1 minute) and at 60 and 120 minutes. The Premature Infant Comfort Scale (PICS) was used to assess comfort, while the Neonatal Stress Scale (NSS) was used to evaluate stress.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — One of the investigators created a randomization sequence using a simple random numbers table and determined the groups. Another researcher assigned premature infants to the study groups according to the order of hospitalization in the unit, and the same researcher also applied the intervention. Thus, each infant experienced all three positions in a crossover design by the end of the study. Infants in all three groups were positioned for two hours in each posture, totaling six hours by the end of the study. Immediately after positioning in each posture, and at 1, 30, 60, 90, and 120 minutes, heart rate and oxygen saturation (SpO₂) values were recorded from bedside monitors, and respiratory rate was counted over one minute. Comfort and stress scores were assessed immediately after positioning (1 minute) and at 60 and 120 minutes. The Premature Infant Comfort Scale (PICS) was used to assess comfort, while the Neonatal Stress Scale (NSS) was used to evaluate stress.
  Other Names: Group 1 (SQP) was positioned in the order: supine (S), quarter prone (Q), and prone (P)

SUMMARY:
A randomized crossover study was made to investigate the effect of different positions on the comfort, stress, and physiological functions of premature infants receiving non-invasive mechanical ventilation in the neonatal intensive care unit (NICU).

DETAILED DESCRIPTION:
Positioning is a crucial care practice for premature infants receiving non-invasive mechanical ventilation, as it creates a safe and confined environment similar to the uterus. In addition to creating a secure environment, positioning supports skin integrity, aids respiratory and circulatory functions , prevents musculoskeletal problems, reduces pain and stress from treatment and care interventions, promotes safe sleep, enhances comfort, and thereby accelerates the recovery process. These practices provide numerous physiological and neurodevelopmental benefits. In premature infants, improper timing and technique in positioning can lead to major risks, including cranial deformities, restricted movement in the arms and legs, postural deformities such as ankle and shoulder extension, hip abduction, skin issues like decubitus ulcers, and respiratory and circulatory problems like venous return disorders, hypoxia, and apnea episodes. In the Neonatal Intensive Care Unit (NICU), positioning management is used to reduce infants' pain or discomfort from medical interventions and environmental stimuli. Maintaining proper posture also helps them cope with stress. Stress can negatively affect neonatal brain development. For patients and premature infants on mechanical ventilation, a nest-like bed can be created using towels, blankets, or similar materials that support a flexed posture and enhance comfort. In 24-hour periods, it is important to change the position regularly, at least every three to four hours. Properly positioning the infant in a flexed posture facilitates self-regulatory movements, such as sucking, bringing hands to the mouth, and moving hands over the eyes. Ensuring the infant's comfort reduces startle responses to harmful stimuli, conserves energy, minimizes stress, and helps maintain physiological balance. Reducing the infant's stress and enhancing comfort through developmental care supports neurodevelopment. Positioning is a non-invasive practice in caring for premature infants and forms a key part of developmentally supportive care.

Nurses should adjust infants' positions according to their unique physiological conditions rather than relying on a single position, aiming to reduce sequelae associated with prolonged hospitalization and to support the infants' growth and recovery. According to researchers' observations and experience, premature infants positioned in quarter prone or stomach positions show better ventilation, better oxygenation, and fewer episodes of apnea. Due to the varying results in the literature, we recognize the need to validate these observations scientifically. The findings are expected to make a valuable contribution to our clinical practices and scientific knowledge in this field.In light of this information, our study aims to investigate the effects of positioning premature infants receiving non-invasive mechanical ventilation in the neonatal intensive care unit in different positions on their comfort, stress levels, and physiological functions (heart rate, SpO₂, and respiratory rate). It was tested the hypotheses that there Positioning premature infants in different positions (supine, prone, and quarter prone) during non-invasive mechanical ventilation in the Neonatal Intensive Care Unit does not affect their comfort levels, stress levels and heart rate, oxygen saturation (SpO₂), or respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* born between 28 and 36 gestational weeks, with no congenital anomalies, no intraventricular hemorrhage or periventricular leukomalacia, and no history of surgical interventions.

Exclusion Criteria:

* - Congenital anomaly,
* Has a clinical, surgical or congenital problem that makes the positions impossible,
* Surgical intervention,
* Intracranial hemorrhage and/or periventricular leukomalacia,
* Bronchopulmonary dysplasia

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
The Premature Infant Comfort after positioning at 1. minutes | After positioning at 1. minutes
  assessed using the The Premature Infant Comfort Scale (PICS).. PICS is a multidimensional scale that assesses comfort and pain behaviorally and physiologically. It is a 5-point Likert-type scale, with each item rated from 1 (poor) to 5 (good). Thus, the highest comfort score is 35, and the lowest is 7. A total score of ≥17 is the threshold for comfort, indicating the need for pain-relieving intervention.
The Premature Infant Comfort after positioning at 60 minutes | After positioning at 60 minutes
  assessed using the The Premature Infant Comfort Scale (PICS).. PICS is a multidimensional scale that assesses comfort and pain behaviorally and physiologically. It is a 5-point Likert-type scale, with each item rated from 1 (poor) to 5 (good). Thus, the highest comfort score is 35, and the lowest is 7. A total score of ≥17 is the threshold for comfort, indicating the need for pain-relieving intervention.
The Premature Infant Comfort after positioning at 120 minutes | After positioning at 120 minutes
  assessed using the Premature Infant Comfort Scale. PICS is a multidimensional scale that assesses comfort and pain behaviorally and physiologically. It is a 5-point Likert-type scale, with each item rated from 1 (poor) to 5 (good). Thus, the highest comfort score is 35, and the lowest is 7. A total score of ≥17 is the threshold for comfort, indicating the need for pain-relieving intervention.
The Neonatal Stress After positioning at 1. minutes | After positioning at 1. minutes
  assessed using the The Neonatal Stress Scale (NSS) was developed to assess stress in premature infants. The scale consists of eight subgroups (facial expression, body color, respiration, activity level, consolability, muscle tone, extremities, and posture) and includes 24 items rated on a 3-point Likert scale. Each subgroup is scored from 0 to 2 points, with a maximum score of 16 and a minimum score of 0. A score of zero indicates no stress, while higher scores indicate increasing stress levels.
The Neonatal Stress After positioning at 60 minutes | After positioning at 60 minutes
  assessed using the The Neonatal Stress Scale (NSS) was developed to assess stress in premature infants. The scale consists of eight subgroups (facial expression, body color, respiration, activity level, consolability, muscle tone, extremities, and posture) and includes 24 items rated on a 3-point Likert scale. Each subgroup is scored from 0 to 2 points, with a maximum score of 16 and a minimum score of 0. A score of zero indicates no stress, while higher scores indicate increasing stress levels.
The Neonatal Stress After positioning at 120 minutes | The Neonatal Stress After positioning at 120 minutes
  assessed using the The Neonatal Stress Scale (NSS) was developed to assess stress in premature infants. The scale consists of eight subgroups (facial expression, body color, respiration, activity level, consolability, muscle tone, extremities, and posture) and includes 24 items rated on a 3-point Likert scale. Each subgroup is scored from 0 to 2 points, with a maximum score of 16 and a minimum score of 0. A score of zero indicates no stress, while higher scores indicate increasing stress levels.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Güler, PhD, Study Chair — Aydin Adnan Menderes University
Locations (2):
- Turkey (Türkiye) (2):
  - Aydın Adnan Menderes University, Aydin
  - Turkey Aydın Adnan Menderes University, Medicine and Health Sciences Research and Applications Hospital, Neonatal Intensive Care Unit, Aydin

IPD SHARING:
Plan to Share IPD: Yes
the data sets generated during and/or analyzed during the current study are available from the correponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request